CLINICAL TRIAL: NCT07019311
Title: Effect of Thera-Band Versus Swiss Ball Exercises on Postural Stability in Post Mastectomy Lymphedema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Afkar Zaki Abdullah Elbanouby, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005215
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Post Mastectomy Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thera-Band exercises + Traditional physical therapy program (Experimental): This group will consist of 32 patients with unilateral lymphedema following mastectomy. Participants will perform Thera-Band resistance exercises in addition to a traditional physical therapy program, 3 times per week for eight consecutive weeks.
  Interventions: Other: Thera-Band exercises; Other: Traditional physical therapy program
- Swiss ball exercises + Traditional physical therapy program (Experimental): This group will consist of 32 patients with unilateral lymphedema following mastectomy. Participants will perform Swiss ball exercises in addition to a traditional physical therapy program, 3 times per week for eight consecutive weeks.
  Interventions: Other: Swiss ball exercises; Other: Traditional physical therapy program

INTERVENTIONS:
Other: Thera-Band exercises — Participants in the first experimental group performed a Thera-Band exercise program 3 sessions weekly, for 8 weeks with progressive resistance, divided into four 2-week phases. Each 60-minute session included a 10-min warm-up (walking, jogging, and calisthenics), 45-min Thera-Band exercises, and 5-min cool-down. Phase 1 focused on major muscle groups (e.g., shoulder press, biceps curl). Phase 2 included trunk and leg-focused moves (e.g., reverse flies, lunge). Phase 3 added advanced resistance (e.g., chest press, deadlift). Phase 4 targeted core and lower body (e.g., diagonal chop, squat). Exercises changed every phase to progressively strengthen different muscle groups.
  Arms: Thera-Band exercises + Traditional physical therapy program
Other: Swiss ball exercises — Participants in the second experimental group performed Swiss ball exercises 3 sessions weekly, for 8 weeks. Exercises included warm-up (15-5 mins), core Swiss ball training (progressing from 1 to 4 sets), and cool-down. Each session focused on abdominal, back, leg, trunk, and balance training using varied exercises performed for 30 seconds with rest. Exercise intensity ranged from 80-95% of max effort, increasing weekly. The Swiss ball size was selected based on patient height to ensure proper posture. Sessions gradually increased in duration and difficulty, ending with breathing and stretching for recovery.
  Arms: Swiss ball exercises + Traditional physical therapy program
Other: Traditional physical therapy program — Participants in both experimental groups performed a traditional physical therapy program in the form of complex decongestive physical therapy(CDPT), including (manual lymphatic drainage, compression, exercise and skin care) and balance training, 3 sessions weekly, for 8 weeks.

SUMMARY:
The purpose of the study is to determine the effect of Thera-band exercises versus Swiss ball exercises on postural stability in unilateral post mastectomy lymphedema.

DETAILED DESCRIPTION:
The need for this study develops from the lack of information in the published studies about the effectiveness of Thera-band exercises and Swiss ball exercise on balance in unilateral post mastectomy lymphedema.

Lymphedema is a chronic and progressive condition associated with functional impairment of the body segment.

The asymmetry between hemi Corp related to the range of motion, muscle strength, sensory stimuli and volume, reduce the ability to perceive and integrate information on the maintenance of the center of gravity and postural balance.

The damage in the balance of patients with breast cancer is pointed out in the literature and is related to factors related to surgical intervention, adjuvant treatment, or even unilateral asymmetry caused by upper limb lymphedema.

Core stability exercises improve neuromuscular system performance that causes the optimal lumbar-pelvic -hip chain mobility and good acceleration and deceleration, appropriate muscular balance, proximal stability and good function.

Progressive resistance training interventions designed to increase strength and reduce the falls in elderly were effective in reducing both rate of falls and risk of falling, especially when some form of balance exercise was an integral part of the program.

The present study is designed to investigate the effect of Thera-band exercises versus Swiss ball exercises on balance in unilateral post mastectomy lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Patients are females.
* Patient with post mastectomy unilateral lymphedema.
* Their age will range from (30-50) years.
* Patients will be given their informed consent.

Exclusion Criteria:

* Musculoskeletal disorders that will impair performance during training and tests.
* Uncontrolled cardiovascular or pulmonary diseases.
* Neurological and renal disorders.
* Metabolic or vascular disease with a neurological component such as diabetes.
* Malignant conditions.
* Primary lymphedema.
* Psychiatric illness, severe behavior or cognitive disorders.
* Uncooperative patients.
* Pregnancy.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-11 (Estimated); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Center of Pressure (COP) | 8 weeks
  The Wii Balance Board (WBB) will be used to measure the Center of Pressure (COP), which represents the point location of the vertical ground reaction force vector. This outcome reflects the user's weight distribution and is a key indicator of balance and postural control. COP will be assessed in both the mediolateral (X-axis: left-right) and anteroposterior (Y-axis: front-back) directions, allowing evaluation of postural sway and dynamic weight shifting during balance tasks.
Total Force (Weight) | 8 weeks
  Total vertical ground reaction force will be calculated by summing the readings from all four pressure sensors on the WBB. This measure provides an estimate of the user's body weight and enables monitoring of force fluctuations during dynamic or static postural tasks, serving as an indirect marker of load-bearing and movement initiation or compensation patterns.
Load Distribution | 8 weeks
  The WBB will quantify the distribution of body weight across the left vs. right and front vs. back regions of the platform. This load distribution outcome helps identify asymmetries in stance or postural alignment, which can be critical in populations with balance deficits or musculoskeletal impairments. The measure allows for detailed analysis of postural strategy and weight-bearing preference.

SECONDARY OUTCOMES:
Limb volume measurement | 8 weeks
  Limb volume will be measured using the truncated cone method with circumferential measurements taken at 10-cm intervals (at 0, 10, 20, 30, and 40 cm from the ulnar styloid). The patient will be seated with the limb supported horizontally on a bedside table. A 1-cm retractable fiberglass tape will be used, and an adhesive measuring strip from axilla to wrist will ensure consistency. Segment volume will be calculated using the formula: V = h × (C1² + C1×C2 + C2²) / (12π), where C1 and C2 are the circumferences and h is the 10 cm distance between them.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Mahmoud Abdelkhalek Khalaf, Study Chair — Professor, Cairo university; Khadra Mohamed Ali, Study Director — Assistant Professor, Cairo university; Eid Rizk El Gammal, Study Director — Assistant Professor, Al-Azhar university
Locations (1):
- Damanhour Oncology Center, Damanhūr, Egypt